CLINICAL TRIAL: NCT03121209
Title: Carotid Revascularization and Medical Management for Asymptomatic Carotid Stenosis Trial - Hemodynamics
Brief Title: Carotid Revascularization and Medical Management for Asymptomatic Carotid Stenosis Trial - Hemodynamics (CREST-H)
Acronym: CREST-H
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Mayo Clinic (Other); University of Alabama at Birmingham (Other); University of Maryland (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Randolph S. Marshall, MD, Professor of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAR5617; 1R01NS097876-01A1 (NIH)
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Internal Carotid Artery Stenosis; Cognitive Impairment
MeSH Terms: conditions — Carotid Stenosis; Cognitive Dysfunction | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Phase 3 prospective blinded outcome randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: single blind by outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Revascularization Arm (CEA or CAS) (Active Comparator): These patients will have been randomized (via the parent trial, CREST-2) to receive intensive medical management as well as either Carotid Endarterectomy (CEA--if they are in the parent study Surgical trial) or Carotid Artery Stenting (CAS--if they are in the parent study Stenting trial).
  Interventions: Procedure: Revascularization
- Intensive Medical Management (IMM) Arm (Active Comparator): These patients will have been randomized (via the parent trial, CREST-2) to receive medical management only, which includes aspirin. high dose cholesterol lowering agent to a target LDL<70, intensive blood pressure management to target <130/80, smoking cessation, and diabetic control.
  Interventions: Other: Intensive Medical Management (IMM) alone

INTERVENTIONS:
Procedure: Revascularization — Patients in this arm are randomized to CEA/CAS plus IMM
  Arms: Revascularization Arm (CEA or CAS)
Other: Intensive Medical Management (IMM) alone — Patients in this arm are randomized to intensive medical management (IMM) alone
  Arms: Intensive Medical Management (IMM) Arm

SUMMARY:
We aim to determine whether cognitive impairment attributable to cerebral hemodynamic impairment in patients with high-grade asymptomatic carotid artery stenosis is reversible with restoration of flow. To accomplish this aim CREST-H will add on to the NINDS-sponsored CREST-2 trial (parallel, outcome-blinded Phase 3 clinical trials for patients with asymptomatic high-grade carotid artery stenosis which will compare carotid endarterectomy plus intensive medical management (IMM) versus IMM alone (n=1,240), and carotid artery stenting plus IMM versus IMM alone (n=1,240) to prevent stroke and death).

CREST-H addresses the intriguing question of whether cognitive impairment can be reversed when it arises from abnormal cerebral hemodynamic perfusion in a hemodynamically impaired subset of the CREST-2 -randomized patients. We will enroll 385 patients from CREST-2, all of whom receive cognitive assessments at baseline and yearly thereafter. We anticipate identifying 100 patients with hemodynamic impairment as measured by an inter-hemispheral MRI perfusion "time to peak" (TTP) delay on the side of stenosis. Among those who are found to be hemodynamically impaired and have baseline cognitive impairment, the cognitive batteries at baseline and at 1 year will determine if those with flow failure who are randomized to a revascularization arm in CREST-2 will have better cognitive outcomes than those in the medical-only arm compared with this treatment difference for those who have no flow failure.

We hypothesize that hemodynamically significant "asymptomatic" carotid disease may represent one of the few examples of treatable causes of cognitive impairment. If cognitive decline can be reversed in these patients, then we will have established a new indication for carotid revascularization independent of the risk of recurrent stroke.

DETAILED DESCRIPTION:
CREST-H sites will be drawn from actively-enrolling CREST-2 centers. The additional information obtained in CREST-H in this protocol will be the MR or CT imaging, which will be done at baseline for all patients enrolled in CREST-H, and at 1 year for those with hemodynamic impairment at baseline. The protocol will recommend an unblinded investigator at each CREST-H site who will order and obtain the study-related MRI sequences, upload de-identified image files to the CREST-2 central imaging site at U Maryland, and maintain blinding of the hemodynamic imaging data for their site (see Blinding below). Image analysis will be done at UCLA (for perfusion studies) and at Mayo Rochester for structural scans -- silent infarcts, WMH and microbleeds. Data management and statistical analysis will be done at UAB, which serves this role for CREST-2.

Cognitive Assessment.

CREST-H will use existing CREST-2 cognitive assessment infrastructure -- the Survey Research Unit at University of Alabama Birmingham. Added to the current CREST-2 battery is the Oral Trail Making A & B as an additional measure of executive function, which will be administered to every CREST-2 patient, regardless of their participation in CREST-H. Cognitive assessments in CREST-H must take place prior to revascularization or within two weeks after assignment to medical therapy alone. Testing in CREST-2 is repeated at 1 year, and every year thereafter up to 4 years. At each test interval, a composite (mean) Z-score is derived from published normative samples for each test outcome. The CREST-H primary outcome will be at 1 year in which the change in the composite Z-score from baseline will be calculated. Covariates will include age, education and depression. The test battery will be administered by a blinded assessor the same way for all CREST-2 and CREST-H enrolled patients. The cognitive domains being assessed in CREST-2/H are entirely consistent with those encompassed within the NINDS Common Data Elements (CDE).

Imaging protocol.

Multimodal MRI or CT perfusion imaging will be performed at baseline on every study subject.

Multimodal MRI, including routine parenchymal sequences and PWI utilizing dynamic susceptibility contrast technique, will be acquired at each participating CREST H site who have been approved for this imaging modality. CT perfusion, using iodinated contrast, will be used as an alternative PWI image for sites approved for this modality. Imaging will take place within 14 days after CREST-H enrollment and prior to any CREST 2 intervention for those randomized to CEA or CAS.

Standardized contrast agent injection protocol, appropriate preparation, and IV setup is used to ensure good scan quality. An antecubital vein IV catheter of 18-20 gauge is required. A test injection will be performed with approximately 10 ml of normal saline solution.

MRI image acquisition DWI/ADC (b=0, 1000 s/mm2 applied in each of three principal gradient directions), FLAIR, high-resolution T1, and GRE sequences will be acquired on 1.5-3.0 T scanners equipped with echo-planar imaging capability, using standard clinical protocols at participating CREST-H sites Total scanning time will be approximately 40 minutes. PWI acquisition protocol will be standardized across all CREST-H sites, using sequential T2*-weighted (gradient echo) EPI time sequence scanning. A modified 2-phase contrast injection scheme will be used to perform CEMRA and DSC perfusion imaging, without need for additional contrast.

CT perfusion imaging will follow the protocol outlined in the updated Imaging MOP for CREST-H. The CT perfusion study is identical to the clinical CTP protocol used for acute stroke imaging in most institutions.

Perfusion imaging analysis.

PWI source images will be sent to the core laboratory at UCLA and processed with the OleaSphere software platform, using deconvolution of tissue and arterial signals in an expedited manner, yielding standardized data regardless of the acquisition system at each site. Hemodynamic impairment is defined as TTP >1.25 sec in the middle cerebral artery and anterior cerebral artery territories of the ipsilateral hemisphere to the carotid lesion compared with the same territory in the opposite hemisphere. Longitudinal analyses will investigate the change in the TTP >1.25 sec lesion at 1 year comparing the revascularization versus the medical only arm. Continuous values for this volumetric change will be used to calculate the correlation between degree of cognitive change and degree of perfusion change. The continuous Tmax variable, as well as standard perfusion parameters of CBV, CBF Tmax, and MTT will be analyzed on the serial imaging studies in each case with MR imaging. Co-registered, voxel-based changes in serial perfusion values will also be explored with multiparametric (e.g. CBV, CBF, Tmax, MTT) values.

Image de-identification and blinding.

All MR or CT image files will be de-identified under the supervision of an unblinded Investigator (UI) at each institution and uploaded to the CREST-2 Imaging Core site at U Maryland. In order to assure that the PWI scan information from CREST-H does not compromise the integrity of the parent trial, the results of the perfusion scan will be blinded to the investigator team.

Image transfer.

Participating sites will utilize the same file transfer protocol (ftp) to transfer images to U Maryland for CREST-H as is already established for CREST-2. The images will be stored in a HIPAA-compliant, firewall protected server within the U Maryland archival system. A CREST-2 dedicated ftp linkage between the VIC at U Maryland and UCLA; and the VIC at U Maryland and Mayo-Rochester will be utilized to make each perfusion image file available for download by UCLA (Liebeskind lab) and each structural image (DWI, FLAIR, GRE) by Mayo-Rochester (Huston lab).

MRI structural analysis.

Structural MRI analysis at Mayo-Rochester will utilize NIH NINDS Common Data Elements developed for the CREST-2 grant. The following definitions apply:

1. silent infarct --- non-confluent hyperintense lesion >1mm on FLAIR sequence on 1-year MRI not present on baseline FLAIR MRI.
2. Cerebral microbleed - hypointense 1-2mm non-confluent lesion on baseline GRE sequence.
3. WMH volume -- White matter hyperintensity volume refers to confluent periventricular high intensity lesions on FLAIR imaging, and will be derived using an automated T2 WMH quantification at the Huston lab.

Data from image analysis (TTP delay, WMHV, silent infarct count, microbleed count) performed at UCLA and Mayo-Rochester will be entered electronically on CREST-H data forms via the CREST-2 SDCC website at UAB, where it will be stored on a separate webpage linked to the rest of the CREST-2 data, including baseline and yearly cognitive assessments. The electronic data entry system (eDES) for CREST-2 is a mature system, successfully reviewed by FDA audit in other studies, providing standard approaches for entry-confirmation-locking of data forms, and supporting range and validity checking for data provided.

. Analysis.

Specific Aim 1. To determine whether cognition can be improved by revascularization among a subset of CREST-2 patients with hemodynamic impairment at baseline.

The primary hypothesis is to assess if the magnitude of the treatment differences (revascularization versus medical management alone) differs between those with flow failure compared to those without flow failure using the Z-scored cognitive outcomes (C0, C(1). That is, the primary hypothesis is an interaction hypothesis that will be assessed using linear regression, specifically: (C1 - C0) = β0 + β1T + β2F + β3TF + β4C0 + (other covariates), where C1 is the cognitive z-score at year 1, C0 the cognitive z-score at baseline, T the treatment indicator variable, F the flow failure indicator variable, and βi the regression parameters to be estimated. The parameter of interest for the primary hypothesis is then β3 that would assess if the magnitude of treatment difference in the change in cognitive score between baseline and 1-year is similar for those with versus without flow failure.

Secondary Aims: To determine if the number of silent infarcts and white matter hyperintensity volume at 1 year is different between the revascularization and the medical-only arms.

For the secondary aims we will calculate the number of new silent cerebral infarctions occurring over the first year, and the change in the WMH volume. The approach for analysis of the number of new silent infarcts will depend on the average number and distribution of the number of new infarcts. The analytic approach will be linear regression if the number of new infarcts is large (considered more likely the case), or Poisson Regression if the number is smaller (considered less likely the case). The analysis of the change in WMH will use a linear regression approach.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled and randomized into CREST-2 (parent study)
* Inclusion criteria for CREST-2
* age 35-86

Exclusion Criteria (in addition to the exclusion criteria for CREST-2):

* unable to undergo MRI (e.g. metal in body, pacemaker)
* known allergy gadolinium contrast dye
* pre-existing diagnosis of dementia
* contralateral ICA stenosis >70% by MRA, CTA or Doppler ultrasound
* history of severe head trauma
* major depression
* education less than 8 years

Ages: 35 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive score at 1 year | 1 year
  Change in composite cognitive Z-score at 1 year will be computed from the cognitive battery of the Carotid Revascularization and Medical Management for Asymptomatic Carotid Stenosis Trial (CREST-2; NCT02089217). Range: -2.0 to 2.0. Positive Z-score change indicates improvement; negative Z-score change indicates worsening.

SECONDARY OUTCOMES:
MRI-determined silent infarcts present at 1 year that were not present at baseline. | 1 year
  A neuroradiology study investigator assesses for new silent infarcts as defined by any non-confluent hyperintense lesion >3mm on T2 FLAIR sequence on 1-year MRI not present on baseline T2 FLAIR MRI
Change from baseline of White matter hyperintensity (WMH) volume as measured by T2 FLAIR sequence on brain MRI. | 1 year
  A neuroradiology study investigator assesses for change in White matter hyperintensity (WMH) volume as defined by confluent periventricular high intensity lesions on T2 Fluid Attenuated Inversion Recovery (FLAIR) imaging.

OTHER OUTCOMES:
Cognitive score beyond 1 year | 2, 3, and 4 years
  Change in composite Z-score from baseline to 2-4 years on the CREST-2 cognitive battery. Range: -2.0 to 2.0. Positive Z-score change indicates improvement; negative Z-score change indicates worsening.
Correlation between change in cognition at 1 year, as measured in Outcome 1, and change in brain blood flow at 1 year as measured by time-to-peak (TTP) perfusion-weighted imaging (PWI) by MRI or computed tomography (CT). | 1 year
  Time-to-peak (TTP) perfusion weighted imaging (PWI) will be derived using a semi-automated software platform that computes quantitative perfusion maps.
Correlation of between change in cognition at 1 year and change in brain blood flow using other MRI PWI markers (CBF, CBV, Tmax). | 1 year
  CBF, CBV, and Tmax will be derived using a semi-automated software platform that computes quantitative perfusion maps.

CONTACTS AND LOCATIONS:
Overall Officials: Randolph S Marshall, MD, Study Chair — Columbia University; Ronald M Lazar, PhD, Study Director — University of Alabama at Birmingham; E Sander Connolly, MD, Study Director — Columbia University; David S Liebeskind, MD, Study Director — University of California, Los Angeles
Locations (58):
- United States (56):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Huntsville Hospital/ Heart Center Research Alabama, Huntsville, Alabama
  - St. Joseph's Hospital and Medical Center/ Barrow, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Keck Medical Center of University of Southern California, Los Angeles, California
  - University of California at Los Angeles, Los Angeles, California
  - Kaiser Permanente, San Diego, California
  - University of California San Diego, San Diego, California
  - San Francisco VA Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - University of Florida Health at Shands, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Mercy Health Riverside, Rockford, Illinois
  - University of Iowa, Iowa City, Iowa
  - Ochsner Health System, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland VA, Baltimore, Maryland
  - Adventist HealthCare/White Oak Medical Center, Gaithersburg, Maryland
  - Michigan Vascular Center/McLaren-Flint, Flint, Michigan
  - Minneapolis Clinic of Neurology, Ltd./ North Memorial Medical Center, Golden Valley, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mercy Hospital St Louis, St Louis, Missouri
  - SUNY Buffalo, Buffalo, New York
  - New York Presbyterian Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Novant Health Forsythe, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State Medical Center, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - UPMC Altoona, Altoona, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian University Hospital, Pittsburgh, Pennsylvania
  - The Miriam Hospital/ Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - North Central Heart Institute, Sioux Falls, South Dakota
  - Tennova Healthcare/ Turkey Creek Medical Center, Knoxville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Health Care, Falls Church, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - University of Washington Medicine-Harborview Medical Center, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
  - Gundersen Clinic, Ltd, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: Yes
To share individual participant data (IPD) of baseline characteristics, follow up, outcomes, etc. based on NIH/NINDS requirements.
Supporting Information: Study Protocol
Time Frame: As per NIH/NINDS requirements.
Access Criteria: All items required by NIH/NINDS will be publicly shared.

REFERENCES:
- [Background] Marshall RS, Lazar RM, Liebeskind DS, Connolly ES, Howard G, Lal BK, Huston J 3rd, Meschia JF, Brott TG. Carotid revascularization and medical management for asymptomatic carotid stenosis - Hemodynamics (CREST-H): Study design and rationale. Int J Stroke. 2018 Dec;13(9):985-991. doi: 10.1177/1747493018790088. Epub 2018 Aug 22. PMID 30132751
- [Background] Marshall RS, Liebeskind DS, Iii JH, Edwards LJ, Howard G, Meschia JF, Brott TG, Lal BK, Heck D, Lanzino G, Sangha N, Kashyap VS, Morales CD, Cotton-Samuel D, Rivera AM, Brickman AM, Lazar RM. Cortical Thinning in High-Grade Asymptomatic Carotid Stenosis. J Stroke. 2023 Jan;25(1):92-100. doi: 10.5853/jos.2022.02285. Epub 2023 Jan 3. PMID 36592969